CLINICAL TRIAL: NCT02561676
Title: Improving Functioning in Persons With Chronic Pain Post-SCI Through Virtual Classroom Education
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: eMindful.com (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-860-14
Record Dates: First submitted 2015-02-11; First posted 2015-09-28 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Chronic Pain; Spinal Cord Injuries
Keywords: Mindfulness; Spinal Cord Injury
MeSH Terms: conditions — Chronic Pain; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-Based Education Program Type 1 (Experimental): The education program involves ten weeks of web-based classes (1.5 hours per class) given once per week with daily homework assignments of approximately 30 minutes per day.
  Interventions: Other: Education Program Type 1
- Web-Based Education Program Type 2 (Experimental): The education program involves ten weeks of web-based classes (1.5 hours per class) given once per week with daily homework assignments of approximately 30 minutes per day.
  Interventions: Other: Education Program Type 2

INTERVENTIONS:
Other: Education Program Type 1 — The classes will discuss topics related to health and functioning of people with spinal cord injury. During these classes, participants will be given information by the class instructor and will also participate in discussions and other learning activities with the rest of the group. Participants will be assigned activities to complete at home for about 30 minutes per day that relate to the topics discussed in class.
  Arms: Web-Based Education Program Type 1
Other: Education Program Type 2 — The classes will discuss topics related to health and functioning of people with spinal cord injury. During these classes, participants will be given information by the class instructor and will also participate in discussions and other learning activities with the rest of the group. Participants will be assigned activities to complete at home for about 30 minutes per day that relate to the topics discussed in class.
  Arms: Web-Based Education Program Type 2

SUMMARY:
Chronic pain (pain that is that is present for a long period of time) is very common among people with spinal cord injury (SCI).

The purpose of this study is to compare how well two different web-based education programs reduce the level to which chronic pain interferes with daily activities and well-being.

DETAILED DESCRIPTION:
Chronic pain (pain that is present for a long period of time) is common among people with spinal cord injury (SCI). The pain is often severe and can affect daily activities. Unfortunately, common treatments such as medications provide incomplete relief from chronic pain. Thus, persons with SCI have to find alternate ways to live a happy, healthy, and productive life, even with some pain.

The purpose of this study is to compare how well two different web-based education programs reduce the level to which chronic pain interferes with daily activities and well-being.

ELIGIBILITY:
Inclusion Criteria:

* SCI for at least one year
* Chronic pain for at least three months that is moderate to severe
* Fluent in English
* Not currently starting a new pain treatment or changing a previous pain treatment

Exclusion Criteria:

* Lack of access to a computer with high-speed internet access, at home or another location
* Cancer or conditions that may worsen over time (such as multiple sclerosis, Parkinson Disease, Alzheimer's disease) and may affect physical or mental functioning
* Significant difficulties with learning or memory
* Previous participation in a health and function education program specifically designed for people with chronic pain and SCI
* Inability to understand English well
* Other conditions not related to SCI that cause pain (such as fibromyalgia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-03; Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in level of pain interference with activities, measured with the Life Interference Subscale of the Multidimensional Pain Inventory (MPI-LIS) | Average of scores obtained during baseline (Week 1 and Week 2) compared to scores obtained during Week 12 (the week in which the program is completed)
  The extent to which pain interferes with daily activities will be measured with the Life Interference Subscale of the Multidimensional Pain Inventory (MPI-LIS). The MPI-LIS is a self-report of extent of interference of pain with life activities and the enjoyment of life. The subscale will be modified to remove two items related to work, as recommended based on a factor analysis of the subscale in persons with SCI.

SECONDARY OUTCOMES:
Change in pain intensity rated on a 0-10 numerical rating scale | Week 12 versus baseline; 3, 6, 12 months post-intervention versus baseline
  Pain intensity will be rated on a 0-10 numerical rating scale (0="no pain" and 10="pain as bad as you can imagine").
Change in Brief Patient Health Questionnaire scores | Week 12 versus baseline; 3, 6, 12 months post-intervention versus baseline
  The Brief Patient Health Questionnaire will be used to assess changes in mental health before and after participation in the education program.
Change in Mental Health Subscale of the SF-36 scores | Week 12 versus baseline; 3, 6, 12 months post-intervention versus baseline
  The Mental Health Subscale of the SF-36 will be used to assess changes in mental health and well-being before and after participation in the education program.
Change in Survey of Pain Attitudes scores | Week 12 versus baseline; 3, 6, 12 months post-intervention versus baseline
  The Survey of Pain Attitudes will be used to assess thoughts and feelings about pain before and after participation in the education program.
Change in Coping Strategies Questionnaire scores | Week 12 versus baseline; 3, 6, 12 months post-intervention versus baseline
  The Coping Strategies Questionnaire will be used to assess thoughts and feelings about pain before and after participation in the education program.
Change in Chronic Pain Acceptance Questionnaire scores | Week 12 versus baseline; 3, 6, 12 months post-intervention versus baseline
  The Chronic Pain Acceptance Questionnaire will be used to assess thoughts and beliefs about pain before and after participation in the education program.
Pain interference with activities, measured with the Life Interference Subscale of the Change in Multidimensional Pain Inventory (MPI-LIS) scores | 3, 6, 12 months post-intervention versus baseline
  The extent to which pain interferes with daily activities will be measured with the Life Interference Subscale of the Multidimensional Pain Inventory (MPI-LIS). The MPI-LIS is a self-report of extent of interference of pain with life activities and the enjoyment of life. The subscale will be modified to remove two items related to work, as recommended based on a factor analysis of the subscale in persons with SCI.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M Zanca, PhD, MPT, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States